CLINICAL TRIAL: NCT05338840
Title: Effects of Mulligan Rotational Movement Versus Medial Gapping Technique on Pain, Range of Motion and Disability in Patients With Knee Osteoarthritis
Brief Title: Mulligan Rotational Movement Versus Medial Gapping Technique in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0142 Iqra
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
Keywords: Mulligan Rotational Movement; Medial Gapping Technique; Pain; Range of Motion; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MULLIGAN (Experimental): ROTATIONAL MOVEMENT
  Interventions: Other: MULLIGAN ROTATIONAL MOVEMENT
- Medial gapping technique (Experimental): Medial gapping technique
  Interventions: Other: Medial gapping technique

INTERVENTIONS:
Other: MULLIGAN ROTATIONAL MOVEMENT — 12 sessions over 6 weeks
  Arms: MULLIGAN
Other: Medial gapping technique — 12 sessions over 6 weeks
  Arms: Medial gapping technique

SUMMARY:
Knee osteoarthritis is a progressive degenerative and non-inflammatory joint disorder. Due to the extensive use and stress placed on knee joint, it is a common site for painful disorders such as knee osteoarthritis. It is seen that medial side of knee is most commonly affected because of weight bearing on medial side. Symptomatically, the knee joint is most commonly affected in osteoarthritis because it requires support, high mobility, and insufficient internal stability. Osteoarthritis of the knee joint affects three parts of the knee joint (medial, lateral, and patellar-femoral joints) and develops slowly, usually over 10-15 years, interfering with daily activities Slow and gentle movements like Tai Chi, Isometric, iso-kinetic and isotonic exercises are considered helpful in increasing joint range of motion and physical function. Stretching and aquatic therapy can also decrease pain and enhance joint flexibility. The aim of this study is to compare the effects of Mulligan rotational movement vs Medial gapping technique on pain, range of motion and disability in knee osteoarthritis.

This study will be a randomized control trial and will be conducted in Riphah clinics and LGH. The study will be completed within the time duration of six months. Non-probability convenient sampling technique will be used to collect the data. Those who will meet the inclusion criteria will be recruited in the group. The sample size of patients with knee osteoarthritis will be taken in this study to find the effects of Mulligan Rotational movements vs. Medial gap technique, aged between 20-40 years, will be allocated to an intervention or control group. The scales used for recording findings will be goniometer, visual analogue scale and modified disability index. Subjects will randomly divide into control group called group A Taking Mulligan therapy and Interventional group called group B taking Median Gapping Technique. 12 sessions over 6 weeks were performed on both groups. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Post-traumatic stiffness of knee
* Restricted range of knee flexion
* Patients with restricted ROM and with Grade 3 or more than three power of knee muscle

Exclusion Criteria:

* Patients with hyper mobile and unstable joints
* Joint infection and loosening,
* Soft tissue injuries around knee joints and
* Other complications of post-fracture

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 6 weeks
  The Numeric pain rating scale is a tool that is used to measure pain.it has a range from 1-10
GONIOMETR | 6 weeks
  Goniometer to measure range of motion. Goniometer is a tool to measure the flexibility of a joint, which is important for injury prevention and execution of many therapeutic movements.
Disability Index Scale | 6 weeks
  Disability Index Scale to measure disability that consist of 10 items, concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lespasio MJ, Piuzzi NS, Husni ME, Muschler GF, Guarino A, Mont MA. Knee Osteoarthritis: A Primer. Perm J. 2017;21:16-183. doi: 10.7812/TPP/16-183. PMID 29035179
- [Background] Lalnunpuii A, Sarkar B, Alam S, Equebal A, Biswas A. Efficacy of mulligan mobilisation as compared to Maitland mobilisation in females with knee osteoarthritis: a double blind randomized controlled trial. International Journal of Therapies and Rehabilitation Research. 2017;6(2):37.
- [Background] Nazir SNB, Rathore FA. Efficacy of Mulligan joint mobilizations and trunk stabilization exercises versus isometric knee strengthening in the management of knee osteoarthritis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2024 May 7;16(1):105. doi: 10.1186/s13102-024-00893-7. PMID 38715135
- [Background] Mehmood Z, Anwar N, Tauqeer S, Shabbir M, Khalid K, Mehmood S. Comparison of Maitland Mobilization and Mulligan Mobilization with Movement in Knee Osteoarthritis Patients. Pakistan Journal of Medical Research. 2021;60(3):126-30
- [Background] Rao RV, Balthillaya G, Prabhu A, Kamath A. Immediate effects of Maitland mobilization versus Mulligan Mobilization with Movement in Osteoarthritis knee- A Randomized Crossover trial. J Bodyw Mov Ther. 2018 Jul;22(3):572-579. doi: 10.1016/j.jbmt.2017.09.017. Epub 2017 Sep 28. PMID 30100279
- [Background] Epskamp S, Dibley H, Ray E, Bond N, White J, Wilkinson A, et al. Range of motion as an outcome measure for knee osteoarthritis interventions in clinical trials: an integrated review. Physical Therapy Reviews. 2020;25(5-6):462-81.